CLINICAL TRIAL: NCT02194712
Title: Detection of Schistosomiasis Circulating Anodic Antigen (CAA) in Travellers After High-risk Water Contact
Brief Title: Detection of Schistosomiasis CAA in Travellers After High-risk Water Contact
Status: Completed | Type: Observational
Sponsor: Meta Roestenberg (Other)
Responsible Party: Sponsor-Investigator, Meta Roestenberg, M.Roestenberg, MD PhD, Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Other Study IDs: CAA48780
Record Dates: First submitted 2014-07-15; First posted 2014-07-18 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Schistosomiasis
Keywords: circulating anodic antigen
MeSH Terms: conditions — Schistosomiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, urine and faeces
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- travellers: travellers with recent (<12 weeks) high risk water contact are included in the study and asked to provide samples for CAA testing
  Interventions: Other: Urine CAA detection

INTERVENTIONS:
Other: Urine CAA detection — In addition to routine diagnostics, serum and urine samples are stored for retrospective UCP-CAA antigen determination.

SUMMARY:
Schistosomiasis is increasingly encountered among travellers returning from the tropics and is known for its focal endemicity, associated with the presence of the snail intermediate host in fresh water. Because schistosomiasis in travellers is often atypical or asymptomatic due to the low intensity of infection, many infections likely go undiagnosed and will develop into chronic schistosomiasis. Conventional treatment of schistosomiasis in travellers with praziquantel 40mg/kg daily dose is known for its modest success rate. Diagnosis of schistosomiasis relies on egg detection, which has a poor sensitivity in low burden infections, or serology, which is inadequate to monitor cure. The department of parasitology of the Leiden University Medical Center has developed a novel diagnostic test based on the up-converting phosphor technology (UCP) to detect circulating anodic antigen (CAA). This test can be performed on serum and urine to detect low intensity schistosomiasis infections and confirm cure after praziquantel treatment. This study will assess the performance of UCP-CAA in travellers with high-risk water contact.

ELIGIBILITY:
Inclusion Criteria:

1. Any self-reported high risk water contact, including wading, showering, surfing, walking along wet shore bare-footed or washing with water from a high-risk source, within 12 weeks prior to reporting to the outpatient department
2. Agreement to perform routine diagnostic procedures to diagnose schistosomiasis infection
3. Willing to provide a maximum of three additional blood samples in addition to routine diagnostic procedures
4. Able to provide informed consent

Exclusion Criteria:

1. Previous treatment for schistosomiasis
2. Known positive schistosomiasis serology
3. The use of immunosuppressive or immunomodulatory drugs at presentation that compromise the interpretation of schistosomiasis serology

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Travellers with reported high-risk water contact <12 weeks before inclusion.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
The sensitivity and specificity of UCP-CAA | 12 weeks after last water contact
  The diagnostic performance of UCP-CAA will be assessed by calculating the sensitivity and specificity of UCP-CAA measurement in travellers 12 weeks after reported high-risk water contact. Routine diagnostics performed by the individual centers, such as serology, will be the standard against which sensitivity (number of cases positive in both tests / number of cases positive in routine diagnostics) and specificity (number of cases negative in both tests / number of cases negative in routine diagnostics) is calculated.

SECONDARY OUTCOMES:
The percentage of travellers with persisting positive UCP-CAA six weeks after conventional praziquantel treatment | six weeks after praziquantel treatment

CONTACTS AND LOCATIONS:
Overall Officials: M.P. Grobusch, Prof. MD. PhD, Principal Investigator — Amsterdam UMC, location VUmc; P.J.J. van Genderen, MD, PhD, Principal Investigator — Harbour Hospital Rotterdam; M. Roestenberg, MD. PhD., Principal Investigator — Leiden University Medical Center
Locations (3):
- Netherlands (3):
  - Academic Medical Center, Amsterdam
  - Leiden University Medical Center, Leiden
  - Harbour Hospital, Rotterdam

REFERENCES:
- [Result] Casacuberta-Partal M, Janse JJ, van Schuijlenburg R, de Vries JJC, Erkens MAA, Suijk K, van Aalst M, Maas JJ, Grobusch MP, van Genderen PJJ, de Dood C, Corstjens PLAM, van Dam GJ, van Lieshout L, Roestenberg M. Antigen-based diagnosis of Schistosoma infection in travellers: a prospective study. J Travel Med. 2020 Jul 14;27(4):taaa055. doi: 10.1093/jtm/taaa055. PMID 32307517